CLINICAL TRIAL: NCT04287140
Title: The Utility of Adding 1 L Intravenous Normal Saline to Standard 75 mg Intramuscular Diclofenac Potassium Injection in Patients Presented to the Emergency Department With an Acute Migraine Attack
Brief Title: The Effect of Intravenous Fluid Therapy in Acute Migraine Attacks
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Haldun Akoglu, Professor of Emergency Medicine, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 09.2019.497
Record Dates: First submitted 2019-12-05; First posted 2020-02-27 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Migraine Disorders; Headache; Acute Pain
Keywords: migraine; pain; normal saline; diclofenac; emergency department; adult; acute attack
MeSH Terms: conditions — Migraine Disorders; Headache; Acute Pain; Pain; Emergencies

STUDY DESIGN:
Intervention Model Description: Allocation: Randomized Intervention Model: Parallel Assignment Masking: Double (Participant, Outcomes Assessor) Primary Purpose: Treatment Secondary Purpose: Adverse Event
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The fluid bag, intravenous pump, serum set will be concealed with opaque coaters, so that patients, doctors, and study investigators will be blinded to the treatment group. Only the nurse who sets the infusion pump will be aware of the treatment group of the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saline (Experimental): 1000 ml of 0.9% normal saline bolus over one hour.
  Interventions: Other: Bolus fluid administration
- No Saline (No Intervention): 10 ml of 0.9% normal saline over one hour.

INTERVENTIONS:
Other: Bolus fluid administration — 1000 ml of 0.9% normal saline bolus over one hour
  Arms: Saline

SUMMARY:
The study is a single-center, double-blind, randomized protocol comparison. The study will be conducted in Marmara University School of Medicine Pendik Training and Research Hospital, Department of Emergency Medicine between April 2020 and October 2020.

The population consists of non-pregnant, adult patients (age of 18 or more) who will be confirmed as migraine according to The International Classification of Headache Disorders 3rd edition (ICHD-3) in the emergency department (ED). After the patient was found suitable for the standard treatment protocol, they will be randomized to receive a 1000 ml bolus of normal saline for 1 hour or normal saline at 10 cc/h for 1 hour. The pain level, functional status, and side effects will be assessed before the beginning, at the 1st hour, 2nd hour and at the 24th hour.

The objective of this study is to determine the effect of an intravenous (IV) fluid bolus on migraine headache among patients treated in the ED.

DETAILED DESCRIPTION:
Introduction Headache is a common complaint that is seen in 70-80% of the population and is a common health problem in emergency services. When evaluating the patient with headache, the first step is to determine whether the headache is primary or secondary (1, 2). Primary headaches are classified according to their symptoms and clinical features. Tension-type headache, migraine, and cluster headache are the most common types of primary headaches (3). Secondary headaches can be classified as headaches due to the head and neck trauma, headaches secondary to neurovascular diseases, and headaches due to withdrawal syndromes secondary to drug abuse (4). Migraine is a primary type of headache characterized by recurrent throbbing (usually unilateral) and associated with photophobia, phonophobia, nausea, and other symptoms. Patients with migraine are usually not pleased with the treatment options due to headaches refractory to treatment (5).

The current approach to the treatment of migraine headaches consists of two components: treatment of the acute migraine attacks, and prophylactic treatment.

According to the World Health Organization (WHO), migraine attacks are the eighth cause of loss of work and performance in the attack period among all lifelong diseases (12). Therefore, effective treatment of migraine attacks is important for the patient and socioeconomic wellbeing of the community. More than 90% of the migraine patients experience acute migraine attacks despite prophylactic treatment and need pain medications (6). Common treatment options used in the ED are phenothiazines (7), serotonin receptor agonists (8), and corticosteroids (9). Headache guideline of the American Academy of Neurology published in 2000 also recommends diclofenac as an effective alternative for the treatment of acute migraine attacks (10, 11). Effective attack therapy has the potential to significantly reduce inefficiency caused by migraine attacks by shortening the duration and reducing the severity of attacks.

Although clinical evidence is uncertain, approximately 40% of patients presenting to the ED with a headache are treated with IV fluids (13). Studies with healthy volunteers showed that mild dehydration reduces the pain threshold and increases central pain-related activity in the anterior cingulate cortex, insula, and thalamus (14). Therefore, it is logical to think that dehydration may trigger acute migraine attacks (15). This led to the common approach to use IV fluids besides pain medications in the ED as a routine procedure. A clear benefit would obviously increase the satisfaction of the patient from the ED services, by increasing the pain threshold, decreasing length of stay, and need for rescue treatment. However, on the contrary, IV fluid therapy without an obvious benefit to the patient has a cost burden on the system, uses labor and time of the ED staff, and may increase the duration of the length of stay in the ED.

Therefore, the aim of this study is to evaluate the efficacy and side effects related to the addition of 1000 cc bolus NS to the standard treatment of migraine in the ED.

ELIGIBILITY:
Inclusion criteria:

* age 18 years or older
* migraine with or without aura according to International Classification of Headache Disorders-3 (ICHD-3) diagnostic criteria confirmed by one-to-one physical exam in the ED
* no declaration and sign of pregnancy, or pregnancy not diagnosed during the ED evaluation before randomization,
* did not receive any IV fluid of 100 cc or more at any facility in the last 12 hours,
* intramuscular diclofenac potassium 75 mg, the standard treatment protocol, is ordered by the physician (no history of known allergic reaction to diclofenac potassium),
* severe dehydration not present as determined by the researcher (hypotension, dry mouth, tongue and eyeballs, decreased urine output)
* no other indication for fluid infusion,
* no contraindication to fluid administration (heart failure patients with diuretic use, renal failure patients with fluid restriction, hemodynamic instability),
* do not have accompanying symptoms and signs related to headaches secondary to other obvious pathologies rather than migraine,
* consent to be included in the study.

Exclusion criteria: no patients will be excluded from the study after randomization. All patients will be evaluated for the primary outcome with an intent-to-treat approach.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
VAS(headache) | at the 2nd hour
  The patient will be asked to place a mark between the 0 and 10 cm points indicated on a 10 cm line, the distance of the marked point to 0 will be taken as the VAS(headache) score in mm.

SECONDARY OUTCOMES:
VAS(headache) | at the 1st hour
  The patient will be asked to place a mark between the 0 and 10 cm points indicated on a 10 cm line, the distance of the marked point to 0 will be taken as the VAS(headache) score in mm.
VAS(nausea) | at the 1st hour
  The patient will be asked to place a mark between the 0 and 10 cm points indicated on a 10 cm line, the distance of the marked point to 0 will be taken as the VASnausea score in mm.
VAS(nausea) | at the 2nd hour
  The patient will be asked to place a mark between the 0 and 10 cm points indicated on a 10 cm line, the distance of the marked point to 0 will be taken as the VASnausea score in mm.
Level of Functional Disability | at the 1st hour
  Categorized as none, mild (makes it difficult to do daily tasks), moderate (not able to do daily tasks), severe (requires bed rest).
Level of Functional Disability | at the 2nd hour
  Categorized as none, mild (makes it difficult to do daily tasks), moderate (not able to do daily tasks), severe (requires bed rest).
Level of Functional Disability | at the 24th hour
  Categorized as none, mild (makes it difficult to do daily tasks), moderate (not able to do daily tasks), severe (requires bed rest).
Adverse Events | at the 1st hour
  The proportion of patients with the following adverse events in each group will be actively pursued during the administration of treatment at the ED: hypernatremia, fluid retention, high blood pressure, injection site reactions
Adverse Events | at the 2nd hour
  The proportion of patients with the following adverse events in each group will be actively pursued during the administration of treatment at the ED: hypernatremia, fluid retention, high blood pressure, injection site reactions
Adverse Events | at the 24th hour
  The proportion of patients with the following adverse events in each group will be actively pursued during the administration of treatment at the ED: hypernatremia, fluid retention, high blood pressure, injection site reactions
Successful Treatment | at the 2nd hour
  The proportion of patients will successful and failed treatments will be compared between study groups. Successful treatment is defined if VAS(headache) is decreased at least 50% from the highest VAS(headache) reported by the patient at any time-point without the need of additional analgesics and/or antiemetics. Failed treatment is defined if VAS(headache) is decreased not more than 10% from the highest VAS(headache) or patient's declaration that the headache is the same at the 2nd hour. All patients defined as failed treatment will be offered the rescue treatment (analgesic and/or antiemetic).
Time-to-discharge | 0 to 24 hours
  Duration between the time of admission to the emergency department and discharge up to 24 hours.
The presence of headache | at the 24th hour
  The patients will be asked to answer if their headache is still present or not, and will be requested to answer as "yes" or "no".
The recurrence of headache | at the 24th hour
  The patients will be asked to answer if their headache has recurred (may still be present or not) or not, and will be requested to answer as "yes" or "no".
Ability to tolerate oral intake | at the 24th hour
  If the patient could eat a regular meal without vomiting in the 30 minutes after intake, they will be considered as "able to eat". All other conditions will be considered a "no".

CONTACTS AND LOCATIONS:
Overall Officials: Haldun Akoglu, MD., Prof., Study Director — Marmara University
Locations (1):
- Marmara University Pendik Education and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Steiner TJ, Stovner LJ, Katsarava Z, Lainez JM, Lampl C, Lanteri-Minet M, Rastenyte D, Ruiz de la Torre E, Tassorelli C, Barre J, Andree C. The impact of headache in Europe: principal results of the Eurolight project. J Headache Pain. 2014 May 21;15(1):31. doi: 10.1186/1129-2377-15-31. PMID 24884549
- [Background] Stovner Lj, Hagen K, Jensen R, Katsarava Z, Lipton R, Scher A, Steiner T, Zwart JA. The global burden of headache: a documentation of headache prevalence and disability worldwide. Cephalalgia. 2007 Mar;27(3):193-210. doi: 10.1111/j.1468-2982.2007.01288.x. PMID 17381554
- [Background] Sharma TL. Common Primary and Secondary Causes of Headache in the Elderly. Headache. 2018 Mar;58(3):479-484. doi: 10.1111/head.13252. Epub 2018 Jan 11. PMID 29322494
- [Background] Lipton RB, Stewart WF, Simon D. Medical consultation for migraine: results from the American Migraine Study. Headache. 1998 Feb;38(2):87-96. doi: 10.1046/j.1526-4610.1998.3802087.x. PMID 9529763
- [Background] Cooke LJ, Becker WJ. Migraine prevalence, treatment and impact: the canadian women and migraine study. Can J Neurol Sci. 2010 Sep;37(5):580-7. doi: 10.1017/s0317167100010738. PMID 21059502
- [Background] Friedman BW, Esses D, Solorzano C, Dua N, Greenwald P, Radulescu R, Chang E, Hochberg M, Campbell C, Aghera A, Valentin T, Paternoster J, Bijur P, Lipton RB, Gallagher EJ. A randomized controlled trial of prochlorperazine versus metoclopramide for treatment of acute migraine. Ann Emerg Med. 2008 Oct;52(4):399-406. doi: 10.1016/j.annemergmed.2007.09.027. Epub 2007 Nov 19. PMID 18006188
- [Background] Bird S, Derry S, Moore RA. Zolmitriptan for acute migraine attacks in adults. Cochrane Database Syst Rev. 2014 May 21;2014(5):CD008616. doi: 10.1002/14651858.CD008616.pub2. PMID 24848613
- [Background] Singh A, Alter HJ, Zaia B. Does the addition of dexamethasone to standard therapy for acute migraine headache decrease the incidence of recurrent headache for patients treated in the emergency department? A meta-analysis and systematic review of the literature. Acad Emerg Med. 2008 Dec;15(12):1223-33. doi: 10.1111/j.1553-2712.2008.00283.x. Epub 2008 Oct 25. PMID 18976336
- [Background] Dahlof C, Bjorkman R. Diclofenac-K (50 and 100 mg) and placebo in the acute treatment of migraine. Cephalalgia. 1993 Apr;13(2):117-23. doi: 10.1046/j.1468-2982.1993.1302117.x. PMID 8495453
- [Background] Massiou H, Serrurier D, Lasserre O, Bousser MG. Effectiveness of oral diclofenac in the acute treatment of common migraine attacks: a double-blind study versus placebo. Cephalalgia. 1991 May;11(2):59-63. doi: 10.1046/j.1468-2982.1991.1102059.x. PMID 1860132
- [Background] Vos T, Flaxman AD, Naghavi M, Lozano R, Michaud C, Ezzati M, Shibuya K, Salomon JA, Abdalla S, Aboyans V, Abraham J, Ackerman I, Aggarwal R, Ahn SY, Ali MK, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Bahalim AN, Barker-Collo S, Barrero LH, Bartels DH, Basanez MG, Baxter A, Bell ML, Benjamin EJ, Bennett D, Bernabe E, Bhalla K, Bhandari B, Bikbov B, Bin Abdulhak A, Birbeck G, Black JA, Blencowe H, Blore JD, Blyth F, Bolliger I, Bonaventure A, Boufous S, Bourne R, Boussinesq M, Braithwaite T, Brayne C, Bridgett L, Brooker S, Brooks P, Brugha TS, Bryan-Hancock C, Bucello C, Buchbinder R, Buckle G, Budke CM, Burch M, Burney P, Burstein R, Calabria B, Campbell B, Canter CE, Carabin H, Carapetis J, Carmona L, Cella C, Charlson F, Chen H, Cheng AT, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahiya M, Dahodwala N, Damsere-Derry J, Danaei G, Davis A, De Leo D, Degenhardt L, Dellavalle R, Delossantos A, Denenberg J, Derrett S, Des Jarlais DC, Dharmaratne SD, Dherani M, Diaz-Torne C, Dolk H, Dorsey ER, Driscoll T, Duber H, Ebel B, Edmond K, Elbaz A, Ali SE, Erskine H, Erwin PJ, Espindola P, Ewoigbokhan SE, Farzadfar F, Feigin V, Felson DT, Ferrari A, Ferri CP, Fevre EM, Finucane MM, Flaxman S, Flood L, Foreman K, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabbe BJ, Gabriel SE, Gakidou E, Ganatra HA, Garcia B, Gaspari F, Gillum RF, Gmel G, Gosselin R, Grainger R, Groeger J, Guillemin F, Gunnell D, Gupta R, Haagsma J, Hagan H, Halasa YA, Hall W, Haring D, Haro JM, Harrison JE, Havmoeller R, Hay RJ, Higashi H, Hill C, Hoen B, Hoffman H, Hotez PJ, Hoy D, Huang JJ, Ibeanusi SE, Jacobsen KH, James SL, Jarvis D, Jasrasaria R, Jayaraman S, Johns N, Jonas JB, Karthikeyan G, Kassebaum N, Kawakami N, Keren A, Khoo JP, King CH, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lalloo R, Laslett LL, Lathlean T, Leasher JL, Lee YY, Leigh J, Lim SS, Limb E, Lin JK, Lipnick M, Lipshultz SE, Liu W, Loane M, Ohno SL, Lyons R, Ma J, Mabweijano J, MacIntyre MF, Malekzadeh R, Mallinger L, Manivannan S, Marcenes W, March L, Margolis DJ, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGill N, McGrath J, Medina-Mora ME, Meltzer M, Mensah GA, Merriman TR, Meyer AC, Miglioli V, Miller M, Miller TR, Mitchell PB, Mocumbi AO, Moffitt TE, Mokdad AA, Monasta L, Montico M, Moradi-Lakeh M, Moran A, Morawska L, Mori R, Murdoch ME, Mwaniki MK, Naidoo K, Nair MN, Naldi L, Narayan KM, Nelson PK, Nelson RG, Nevitt MC, Newton CR, Nolte S, Norman P, Norman R, O'Donnell M, O'Hanlon S, Olives C, Omer SB, Ortblad K, Osborne R, Ozgediz D, Page A, Pahari B, Pandian JD, Rivero AP, Patten SB, Pearce N, Padilla RP, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Phillips MR, Pierce K, Pion S, Polanczyk GV, Polinder S, Pope CA 3rd, Popova S, Porrini E, Pourmalek F, Prince M, Pullan RL, Ramaiah KD, Ranganathan D, Razavi H, Regan M, Rehm JT, Rein DB, Remuzzi G, Richardson K, Rivara FP, Roberts T, Robinson C, De Leon FR, Ronfani L, Room R, Rosenfeld LC, Rushton L, Sacco RL, Saha S, Sampson U, Sanchez-Riera L, Sanman E, Schwebel DC, Scott JG, Segui-Gomez M, Shahraz S, Shepard DS, Shin H, Shivakoti R, Singh D, Singh GM, Singh JA, Singleton J, Sleet DA, Sliwa K, Smith E, Smith JL, Stapelberg NJ, Steer A, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Syed S, Tamburlini G, Tavakkoli M, Taylor HR, Taylor JA, Taylor WJ, Thomas B, Thomson WM, Thurston GD, Tleyjeh IM, Tonelli M, Towbin JA, Truelsen T, Tsilimbaris MK, Ubeda C, Undurraga EA, van der Werf MJ, van Os J, Vavilala MS, Venketasubramanian N, Wang M, Wang W, Watt K, Weatherall DJ, Weinstock MA, Weintraub R, Weisskopf MG, Weissman MM, White RA, Whiteford H, Wiersma ST, Wilkinson JD, Williams HC, Williams SR, Witt E, Wolfe F, Woolf AD, Wulf S, Yeh PH, Zaidi AK, Zheng ZJ, Zonies D, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Years lived with disability (YLDs) for 1160 sequelae of 289 diseases and injuries 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2163-96. doi: 10.1016/S0140-6736(12)61729-2. PMID 23245607
- [Background] Jones CW, Gaughan JP, McLean SA. Epidemiology of intravenous fluid use for headache treatment: Findings from the National Hospital Ambulatory Medical Care Survey. Am J Emerg Med. 2017 May;35(5):778-781. doi: 10.1016/j.ajem.2017.01.030. Epub 2017 Jan 15. PMID 28233646
- [Background] Ogino Y, Kakeda T, Nakamura K, Saito S. Dehydration enhances pain-evoked activation in the human brain compared with rehydration. Anesth Analg. 2014 Jun;118(6):1317-25. doi: 10.1213/ANE.0b013e3182a9b028. PMID 24384865
- [Background] Blau JN. Water deprivation: a new migraine precipitant. Headache. 2005 Jun;45(6):757-9. doi: 10.1111/j.1526-4610.2005.05143_3.x. PMID 15953311